CLINICAL TRIAL: NCT03226691
Title: Peripheral Blood Stem Cell Collection for Sickle Cell Disease (SCD) Patients Using Plerixafor
Brief Title: Peripheral Blood Stem Cell Collection for Sickle Cell Disease (SCD) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 170124; 17-H-0124
Record Dates: First submitted 2017-07-21; First posted 2017-07-24 (Actual); Results first posted 2020-04-20 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2019-06-06

CONDITIONS: Sickle Cell Disease
Keywords: Plerixafor; Leukapheresis; Mobilization; Stem Cells; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — plerixafor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Cohort - Plerixafor (Experimental): Plerixafor at a single dose of 240 microgram/kg
  Interventions: Drug: Plerixafor

INTERVENTIONS:
Drug: Plerixafor — Single-dose subcutaneous administration of plerixafor (Mozobil®) at 240 μg/kg
  Other Names: Mozobil®

SUMMARY:
The constitution of blood relies upon hematopoietic stem cells (HSCs), which stay in the bone marrow and differentiate to all lineages of peripheral blood cells. HSC transplantation is the only curative option currently available for sickle cell disease (SCD) patients either via allogeneic HSC transplantation or HSC-targeted gene therapy. Granulocyte-colony stimulating factor (G-CSF)- mobilized HSCs are frequently utilized in the adult setting of HSC transplantation because of the faster hematologic recovery as compared to bone marrow. As an autologous HSC source for gene therapy, bone marrow harvest has been generally employed since G-CSF has been prohibitive in SCD patients due to granulocyte stimulation and the associated reports of vaso-occlusive crises, multi-organ failure, and death. However, when bone marrow harvest is used, the amounts of collected cells are limited and anesthesia is required. In order to obtain HSCs in large numbers without anesthesia, patients will undergo mobilization followed by large volume apheresis. Plerixafor is an alternative treatment for mobilization without direct stimulation to granulocytes, and it is theoretically applicable for SCD patients. The primary endpoint of this study is to obtain sufficient amounts of HSCs collected from the peripheral blood in SCD patients after plerixafor

mobilization with an acceptable safety profile. The harvested products will be stored as backup for patients undergoing gene therapy as well as allogeneic HSC transplantation.

DETAILED DESCRIPTION:
The constitution of blood relies upon hematopoietic stem cells (HSCs), which stay in the bone marrow and differentiate to all lineages of peripheral blood cells. HSC transplantation is the only curative option currently available for sickle cell disease (SCD) patients either via allogeneic HSC transplantation or HSC-targeted gene therapy. Granulocyte-colony stimulating factor (G-CSF)- mobilized HSCs are frequently utilized in the adult setting of HSC transplantation because of the faster hematologic recovery as compared to bone marrow. As an autologous HSC source for gene therapy, bone marrow harvest has been generally employed since G-CSF has been prohibitive in SCD patients due to granulocyte stimulation and the associated reports of vaso-occlusive crises, multi-organ failure, and death. However, when bone marrow harvest is used, the amounts of collected cells are limited and anesthesia is required. In order to obtain HSCs in large numbers without anesthesia, patients will undergo mobilization followed by large volume apheresis. Plerixafor is an alternative treatment for mobilization without direct stimulation to granulocytes, and it is theoretically applicable for SCD patients. The primary endpoint of this study is to obtain sufficient amounts of HSCs collected from the peripheral blood in SCD patients after plerixafor mobilization with an acceptable safety profile. The harvested products will be stored as backup for patients undergoing gene therapy as well as allogeneic HSC transplantation.

ELIGIBILITY:
* INCLUSION CRITERIA:
* SCD patients who are 18 or older, and (a) planned to enroll in an active allogeneic HSCT study where back-up autologous HSCs are needed; OR (b) are eligible for an allogeneic HSCT study (i.e. have the same disease severity as group (a), but no active allogeneic HSCT study is available), and are willing to donate autologous HSCs for a future gene therapy, gene editing, or allogeneic HSCT study.
* Adequate renal function: serum/plasma creatinine <1.5 mg/dL.
* Adequate liver function: direct bilirubin and ALT <5 times the upper limit of normal range.
* Blood counts: WBC >3,000/mm^3, granulocytes >1,000/mm^3, hemoglobin>7.0g/dL, platelets>150,000/mm^3.
* Female patients of childbearing age should have a negative serum pregnancy test within one week of beginning plerixafor administration, have had a hysterectomy, post-menopausal, or absence of a menses for over a year.
* Meets NIH Department of Transfusion Medicine (DTM) eligibility criteria for blood component donation for in vitro research use (negative serologic tests for syphilis, hepatitis B and C, HIV, and HTLV-1).
* Ability to give informed consent to participate in the protocol.
* Female and male individuals of reproductive potential must agree to one of the contraceptive regimens stated above if sexually active

EXCLUSION CRITERIA:

* Pregnancy. Female patients of childbearing age should have a negative serum pregnancy test within one week of beginning plerixafor administration, except those that have had a hysterectomy, post-menopausal, or an absence of a menses for over a year.
* Active viral, bacterial, fungal, or parasitic infection.
* History of cancer, excluding squamous carcinoma of the skin and cervical carcinoma in situ.
* Active and painful splenomegaly or splenomegaly (size greater than upper limit of normal) determined by ultrasound.
* Allergy to plerixafor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John F Tisdale, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Leonard A, Sharma A, Uchida N, Stroncek D, Panch SR, West K, Molloy E, Hughes TE, Hauffe S, Taylor T, Fitzhugh C, Hankins JS, Wilson M, Tsai SQ, Weiss MJ, Hsieh M, Tisdale JF. Disease severity impacts plerixafor-mobilized stem cell collection in patients with sickle cell disease. Blood Adv. 2021 May 11;5(9):2403-2411. doi: 10.1182/bloodadvances.2021004232. PMID 33956057
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-H-0124.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Plerixafor: Plerixafor at a single dose of 240 microgram/kg
Period: Overall Study
Arm/Group | Experimental: Plerixafor
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: Plerixafor
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sufficient Collection of Hemopoietic Stem Cells (HSCs) Without Serious Adverse Events
Description: Sufficient collection of HSCs (target 2.0x106 CD34+ cells/kg) from the PB after plerixafor mobilization without serious adverse events (SAEs)
Time Frame: 1 day
Population: Individuals with SCD age 18 or greater and are willing to donate HSC collection for future gene therapy or gene editing study, if no allogeneic HSC transplantation study was currently available
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Plerixafor
Number analyzed (Participants) | 15
Participants | 14

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | Experimental: Plerixafor
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Plerixafor (N=15)
Hemolysis (Blood and lymphatic system disorders) | 1
Pain (General disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Plerixafor (N=15)
Anemia (Blood and lymphatic system disorders) | 1
Cardiac disorders - Other specify: irregular heart rate (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Blurred vision (Eye disorders) | 1
Eye disorders - Other specify: double vision (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Bloating (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Edema face (General disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 4
Fever (General disorders) | 1
General disorders and administration site conditions - Other specify: Leg pain (General disorders) | 1
General disorders and administration site conditions - Other specify: Pain (General disorders) | 1
Pain at the subcutaneous port site (General disorders) | 1
Injection site reaction (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 6
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Brachial plexopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 6
Paresthesia (Nervous system disorders) | 6
Spasticity (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Swelling soft tissue left hand, dorsal interspace between thumb and index finger (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT03226691/Prot_SAP_001.pdf